CLINICAL TRIAL: NCT00787150
Title: A Phase 2b, Randomized, Partially Blind (Open Label Warfarin), Active-Controlled (Warfarin), Multicenter Study, To Evaluate The Safety And Efficacy In 2 Doses Of Apixaban In Comparison To Warfarin, Administered For 12 Weeks In Subjects With NVAF
Brief Title: A Phase 2 Study To Evaluate The Safety Of Apixaban In Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0661003
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Warfarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Apixaban 5mg BID (Experimental)
  Interventions: Drug: Apixaban
- Apixaban 2.5mg BID (Experimental)
  Interventions: Drug: Apixaban
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin sodium

INTERVENTIONS:
Drug: Apixaban — Apixaban 5 mg tablet BID for 12 weeks
  Arms: Apixaban 5mg BID
Drug: Apixaban — Apixaban 2.5 mg tablet BID for 12 weeks
  Arms: Apixaban 2.5mg BID
Drug: Warfarin sodium — At each visit, the subject to take appropriate Warfarin tablet (on investigator's order) once a day every morning for 12 weeks
  Arms: Warfarin

SUMMARY:
To assess the effect of two doses of Apixaban (2.5 mg BID and 5 mg BID) versus Warfarin on the composite endpoint of major and clinically relevant non-major bleeding during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years outpatient (regardless of sex)
* Patients diagnosed as non-valvular atrial fibrillation (NVAF)
* One or more following risks of stroke.

Exclusion Criteria:

* Recent cerebral infarction (includes TIA) within 4 weeks of week 0.
* Subjects who have or are suspected to have a serious/hereditary bleeding tendency, such as disseminated intravascular coagulation syndrome (DIC), congenital platelet dysfunction and von Willebrand disease (those suspected from the family history are included).
* Subjects who have or are suspected to have a serious/hereditary thrombogenic tendency (those suspected from the family history are included) or those who require continuation of the Warfarin therapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Japan (18):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Seto, Aichi-ken
  - Pfizer Investigational Site, Touon, Ehime
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kitakyushu, Fukuoka
  - Pfizer Investigational Site, Ōgaki, Gifu
  - Pfizer Investigational Site, Isesaki, Gunma
  - Pfizer Investigational Site, Shibukawa, Gunma
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Higashiibaraki-gunn Ibarakimachi, Ibaraki
  - Pfizer Investigational Site, Zentsujichó, Kagawa-ken
  - Pfizer Investigational Site, Kawasaki, Kanagawa
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo
  - Pfizer Investigational Site, Iwakuni, Yamaguchi

REFERENCES:
- [Derived] Ogawa S, Shinohara Y, Kanmuri K. Safety and efficacy of the oral direct factor xa inhibitor apixaban in Japanese patients with non-valvular atrial fibrillation. -The ARISTOTLE-J study-. Circ J. 2011;75(8):1852-9. doi: 10.1253/circj.cj-10-1183. Epub 2011 Jun 14. PMID 21670542
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661003&StudyName=A%20Phase%202%20Study%20To%20Evaluate%20The%20Safety%20Of%20Apixaban%20In%20Atrial%20Fibrillation

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin: The appropriate dose of warfarin sodium, as 2 mg tablet, to achieve the target prothrombin time - international normalization ratio (PT-INR: 2.0-3.0 for under 70 years old; 2.0-2.6 for 70 years or older) was administered once a day every morning after meal for 12 weeks.
- Apixaban 2.5mg BID: One apixaban 2.5 mg tablet and 1 apixaban 5.0 mg placebo tablet were administered twice a day (morning and evening) after a meal for 12 weeks.
- Apixaban 5.0 mg BID: One apixaban 5.0 mg tablet and 1 apixaban 2.5 mg placebo tablet were administered twice a day (morning and evening) after a meal for 12 weeks.
Period: Overall Study
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Started | 75 (Of 222 participants enrolled 4 discontinued before dosing, made a total of 218 participants started.) | 72 (Of 222 participants enrolled 4 discontinued before dosing, made a total of 218 participants started.) | 71 (Of 222 participants enrolled 4 discontinued before dosing, made a total of 218 participants started.)
Completed | 66 | 65 | 66
Not Completed | 9 | 7 | 5
Not completed — Adverse Event | 4 | 4 | 4
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Dosing incorrect study durg | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID | Total
Number analyzed (Participants) | 74 | 74 | 74 | 222
Age Continuous [Mean (Standard Deviation); unit: years] | 71.7 (7.0) | 69.3 (8.4) | 70.0 (8.1) | 70.3 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 13 | 38
  Male | 60 | 63 | 61 | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major (Per International Society on Thrombosis and Haemostasis [ISTH] Criteria) or Clinically Relevant Non-major Bleeding Adjudicated by Clinical Event Committee During the Treatment Period
Description: Major bleeding event was acute clinically overt bleeding accompanied by decrease in hemoglobin of 2 g/dL or more over a 24-hour period, transfusion of 2 or more units of packed red blood cells, or bleeding that occurs in critical site (e.g., intracranial). Fatal bleeding was also major bleeding event. Clinical relevant non-major bleeding was acute or sub-acute clinically overt bleeding that does not satisfy the criteria for major bleeding and that leads to either hospital admission for bleeding, physician guided medical or surgical treatment for bleeding or a change in antithrombotic therapy.
Time Frame: Baseline to Week 12
Population: The safety analysis set consisted of all treated participants. Two participants (1 each in the apixaban 2.5 mg BID group and apixaban 5.0 mg BID group) were mistakenly administered warfarin and therefore, included in the warfarin group per the statistical analysis plan.
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
participants | 4 | 1 | 1

2. Secondary Outcome: Number of Participants With Total Bleeding Events During the Treatment Period
Description: Total bleeding events consisted of major (per International Society on Thrombosis and Haemostasis [ISTH] Criteria), clinically relevant non-major and minor bleeding events. All acute clinically overt bleeding events not meeting the criteria for either major bleeding or clinically relevant non-major bleeding were classified as minor bleeding.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
participants | 13 | 9 | 17

3. Secondary Outcome: Number of Participants With Major (Per International Society on Thrombosis and Haemostasis [ISTH] Criteria) Bleeding Events During the Treatment Period
Description: Major bleeding event is acute clinically overt bleeding accompanied by decrease in hemoglobin of 2 g/dL or more over a 24-hour period, transfusion of 2 or more units of packed red blood cells, or bleeding that occurs in critical site (e.g., intracranial). Fatal bleeding is also major bleeding event.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
participants | 1 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Relevant Non-major Bleeding Events During the Treatment Period
Description: Clinical relevant non-major bleeding was acute or sub-acute clinically overt bleeding that does not satisfy the criteria for major bleeding and that leads to either hospital admission for bleeding, physician guided medical or surgical treatment for bleeding or a change in antithrombotic therapy.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
participants | 3 | 1 | 1

5. Secondary Outcome: Number of Participants With Stroke or Systemic Embolism During the Intended Treatment Period
Description: The definition of the "Intended Treatment Period" was the period starting on the day of randomization and ending at the later one of either 2 days after the last dose of the study drug or Day 85/Week 12 after the randomization day.
Time Frame: Baseline to Week 12
Population: Full analysis set (FAS) was defined as all randomized participants. Participants were categorized to the group to which they were assigned by the randomization system, regardless of the treatment actually received.
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 74 | 74 | 74
participants | 3 | 0 | 0

6. Secondary Outcome: Number of Participants With Stroke, Systemic Embolism, or All-Cause Death During the Intended Treatment Period
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 74 | 74 | 74
participants | 3 | 0 | 0

7. Secondary Outcome: Number of Participants With Myocardial Infarction or All-Cause Death During the Intended Treatment Period
Description: as for outcome 5
Time Frame: Baseline to Week 12
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 74 | 74 | 74
participants | 0 | 0 | 0

8. Other Pre Specified Outcome: Mean Plasma Apixaban Concentration at Each Time Point in Participants Treated With Apixaban
Description: Sample at 4 hours postdose was to be taken if possible.
Time Frame: 0, 2, 4 hours postdose at Week 1 and Week 8
Population: The pharmacokinetic analysis set was defined as participants treated with apixaban, who were not assessed as major protocol violators, and in whom at least one observation of plasma apixaban concentration. n=number of participants with evaluable data in Apixaban 2.5 mg BID, Apixaban 5.0 mg BID, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 72 | 71
ng/mL
  0 hour post dose at Week 1 (n=68, 70) | 53.31 (28.55) | 119.34 (50.83)
  2 hours post dose at Week 1 (n=68, 70) | 99.43 (44.65) | 201.80 (95.58)
  4 hours post dose at Week 1 (n=38, 35) | 104.09 (44.48) | 224.40 (77.06)
  0 hour post dose at Week 8 (n=67, 66) | 62.83 (37.27) | 137.79 (54.91)
  2 hours post dose at Week 8 (n=67, 66) | 120.16 (57.79) | 250.53 (81.35)
  4 hours post dose at Week 8 (n=35, 29) | 110.58 (49.96) | 244.55 (84.27)

9. Other Pre Specified Outcome: Mean Prothrombin Time (PT) at Each Time Point in Participants Treated With Apixaban
Description: Sample at 4 hours postdose was to be taken if possible.
Time Frame: Week 0, 0, 2, 4 hours postdose at Week 1 and Week 8
Population: The analysis set was based on all participants with relevant measurements. Participants were categorized to the actual treatment received. n=number of subjects with evaluable data in Apixaban 2.5 mg BID, Apixaban 5.0 mg BID, respectively.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 72 | 71
second
  Week 0 (n=72, 71) | 14.54 (2.20) | 14.41 (2.06)
  0 hour post dose at Week 1 (n=67, 70) | 12.22 (1.56) | 12.54 (0.79)
  2 hours post dose at Week 1 (n=68, 70) | 12.46 (0.72) | 13.28 (1.05)
  4 hours post dose at Week 1 (n=38, 35) | 12.36 (0.67) | 13.48 (0.82)
  0 hour post dose at Week 8 (n=67, 66) | 12.09 (0.73) | 12.74 (0.87)
  2 hours post dose at Week 8 (n=67, 66) | 12.68 (0.82) | 13.83 (1.03)
  4 hours post dose at Week 8 (n=35, 29) | 12.47 (0.75) | 13.85 (1.07)

10. Other Pre Specified Outcome: Mean Prothrombin Time-International Normalized Ratio (PT-INR) at Each Time Point in Participants Treated With Apixaban
Description: Blood sample at 4 hours postdose was collected if possible. PT-INR is a standardized measure derived from prothrombin time (PT). The systematic variations in PT assay results are corrected in PT-INR in order to optimize measurements of vitamin K antagonists.
Time Frame: Week 0, 0, 2, 4 hours postdose at Week 1 and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: International normalized ratio
Arm/Group | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 72 | 71
International normalized ratio
  Week 0 (n=72, 71) | 1.76 (0.46) | 1.72 (0.43)
  0 hour post dose at Week 1 (n=67, 70) | 1.30 (0.37) | 1.34 (0.15)
  2 hours post dose at Week 1 (n=68, 70) | 1.33 (0.14) | 1.48 (0.21)
  4 hours post dose at Week 1 (n=38, 35) | 1.30 (0.12) | 1.51 (0.18)
  0 hour post dose at Week 8 (n=67, 66) | 1.27 (0.14) | 1.38 (0.17)
  2 hours post dose at Week 8 (n=67, 66) | 1.37 (0.16) | 1.61 (0.20)
  4 hours post dose at Week 8 (n=35, 29) | 1.34 (0.15) | 1.59 (0.22)

11. Other Pre Specified Outcome: Mean Activated Partial Thromboplastin Time (aPTT) at Each Time Point in Participants Treated With Apixaban
Description: Blood Sample at 4 hours postdose was collected if possible. The aPTT is a screening test for the intrinsic pathway and is sensitive for deficiencies of Factors I, II, V, VIII, IX, X, XI and XII. Higher values than the baseline indicate anticoagulant effects.
Time Frame: Week 0, 0, 2, 4 hours postdose at Week 1 and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Second
Arm/Group | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 72 | 71
Second
  Week 0 (n=72, 71) | 34.51 (5.05) | 32.98 (4.39)
  0 hour post dose at Week 1 (n=67, 70) | 33.26 (10.24) | 33.24 (4.28)
  2 hours post dose at Week 1 (n=68, 70) | 33.04 (3.57) | 35.19 (4.42)
  4 hours oist dose at Week 1 (n=38, 35) | 32.00 (3.49) | 35.36 (5.44)
  0 hour post dose at Week 8 (n=67, 66) | 33.83 (5.18) | 35.65 (4.32)
  2 hours post dose at Week 8 (n=67, 66) | 34.67 (4.39) | 37.92 (4.78)
  4 hours post dose at Week 8 (n=35, 29) | 32.75 (3.86) | 36.46 (5.19)

12. Other Pre Specified Outcome: Mean Anti-Xa Activity (Apixaban Units) at Each Time Point in Participants Treated With Apixaban
Description: Blood sample at 4 hours postdose was collected if possible. Below the limit of quantification (BLQ) was assigned the value 0 for calculation. If 50% or more of the data was BLQ, statistics was not be calculated. Therefore, 0 means not calculated.
Time Frame: Week 0, 0, 2, 4 hours postdose at Week 1 and Week 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 72 | 71
ng/mL
  Week 0 (n=72, 71) | 0 (0) | 0 (0)
  0 hour post dose at Week 1 (n=68, 69) | 45.29 (26.77) | 111.19 (49.02)
  2 hours post dose at Week 1 (n=68, 70) | 94.90 (45.23) | 187.58 (85.72)
  4 hours post dose at Week 1 (n=38, 35) | 99.07 (44.46) | 213.24 (67.54)
  0 hour post dose at Week 8 (n=67, 65) | 56.81 (37.34) | 130.12 (52.20)
  2 hours post dose at Week 8 (n=67, 66) | 114.97 (56.25) | 236.36 (88.08)
  4 hours post dose at Week 8 (n=35, 29) | 103.61 (44.54) | 237.78 (78.58)

13. Other Pre Specified Outcome: Mean Prothrombin Fragment 1+2 (F1+2) at Each Time Point in Participants Treated With Warfarin or Apixaban
Description: Below the limit of quantification (BLQ) was assigned the value 0 for calculation. If 50% or more of the data was BLQ, statistics was not calculated. Therefore, 0 indicates not calculated.
Time Frame: Week 0, Week 1, Week 8
Population: The analysis set was based on all participants with relevant measurements. Participants were categorized to the actual treatment received. n=number of subjects with evaluable data in Warfarin, Apixaban 2.5 mg BID, Apixaban 5.0 mg BID, respectively.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
pmol/L
  Week 0 (n=75, 72, 71) | 144.0 (345.2) | 0 (0) | 91.4 (115.3)
  Week 1 (n=75, 68, 70) | 100.4 (139.0) | 133.8 (105.5) | 137.0 (255.5)
  Week 8 (n=68, 67, 66) | 0 (0) | 152.9 (79.7) | 121.1 (56.3)

14. Other Pre Specified Outcome: Mean D-Dimer at Each Time Point in Participants Treated With Warfarin or Apixaban
Description: Below the limit of quantification (BLQ) was assigned the value 0 for calculation.
Time Frame: Week 0, Week 1, Week 8
Population: The analysis set was based on all participants with relevant measurements. Participants were categorized to the actual treatment received. n=number of participants with evaluable data in Warfarin, Apixaban 2.5 mg BID, Apixaban 5.0 mg BID, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Number analyzed (Participants) | 75 | 72 | 71
ng/mL
  Week 0 (n=75, 72, 71) | 240.4 (333.5) | 297.8 (634.6) | 196.4 (181.4)
  Week 1 (n=75, 68, 70) | 245.2 (325.7) | 209.9 (202.6) | 237.0 (314.3)
  Week 8 (n=68, 67, 66) | 209.9 (201.1) | 227.0 (253.5) | 203.5 (190.6)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Warfarin | Apixaban 2.5mg BID | Apixaban 5.0 mg BID
Serious Adverse Events (participants affected / at risk) | 4/75 | 1/72 | 5/71
Other Adverse Events (participants affected / at risk) | 17/75 | 24/72 | 22/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=75) | Apixaban 2.5mg BID (N=72) | Apixaban 5.0 mg BID (N=71)
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin (N=75) | Apixaban 2.5mg BID (N=72) | Apixaban 5.0 mg BID (N=71)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Fatigue (General disorders) | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 7 | 8 | 8
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 2 | 1
Blood creatine phophkinase increased (Investigations) | 0 | 2 | 2
Blood urine present (Investigations) | 4 | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Blood pressure inadequately controlled (Vascular disorders) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.